CLINICAL TRIAL: NCT07256977
Title: A Multicenter Non-inferiority Randomized Controlled Trial on Minimally Invasive Radical Hysterectomy Using an Endoscopic Stapler to Prevent Tumor Spillage in Stage IB2-IIA1 Cervical Cancer
Brief Title: Minimally Invasive Radical Hysterectomy Using Endoscopic Stapler in Stage IB2 or IIA1 Cervical Cancer
Acronym: SOLUTION2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ajou University School of Medicine (Other); SMG-SNU Boramae Medical Center (Other); Konkuk University (Other); DongGuk University (Other); Keimyung University (Other); National Cancer Center, Korea (Other Government); The Catholic University of Korea (Other); Wonju Severance Christian Hospital (Other); Kangbuk Samsung Hospital (Other); Asan Medical Center (Other); Samsung Medical Center (Other); Sinchon Severance Hospital, Yonsei University College of Medicine (Unknown)
Responsible Party: Principal Investigator, Hee Seung Kim, Clinical Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOLUTION2; 0620202330 (Other Grant/Funding Number: Johnson @ Johnson)
Record Dates: First submitted 2025-10-06; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Cervical Cancer Stage IB2; Cervical Cancer Stage IIa
Keywords: Cervical cancer; open radical hysterectomy; minimally invasive radical hysterectomy; endoscopic stapler; survival; complications; perioperative outcomes; postoperative pain; quality of life; recurrence pattern
MeSH Terms: conditions — Uterine Cervical Neoplasms; Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Open radical hysterectomy (Experimental): Radical hysterectomy is performed via open surgery
  Interventions: Device: Open radical hysterectomy
- Minimally invasive radical hysterectomy (Experimental): Radical hysterectomy is performed via minimally invasive surgery
  Interventions: Device: Minimally invasive radical hysterectomy

INTERVENTIONS:
Device: Open radical hysterectomy — Radical hysterectomy is performed via open surgery, and Wertheim clamp is used for preventing tumor spillage during colpotomy
  Arms: Open radical hysterectomy
Device: Minimally invasive radical hysterectomy — Radical hysterectomy is performed via minimally invasive surgery, and an endoscopic stapler is used for preventing tumor spillage during colpotomy
  Arms: Minimally invasive radical hysterectomy

SUMMARY:
This study is a multicenter, open-label, non-inferiority, randomized controlled, investigator-initiated clinical trial comparing the efficacy and safety of open radical hysterectomy versus minimally invasive radical hysterectomy using an endoscopic stapler as surgical treatments for early cervical cancer.

DETAILED DESCRIPTION:
This study exclusively includes patients with stage IB2 or IIA1 cervical cancer who have tumors measuring 2 cm or larger but less than 4 cm. After randomization, one group undergoes radical hysterectomy via open surgery, while the other group undergoes minimally invasive radical hysterectomy using an endoscopic stapler. This approach using an endoscopic stapler aims to prevent intraoperative exposure of tumor cells to the abdominal cavity, comparable to open surgery, thereby enabling a comparison of therapeutic efficacy and safety.

ELIGIBILITY:
I. Inclusion Criteria:

1. 2018 FIGO stage IB2 or IIA1 cervical cancer (tumor maximum diameter ≥2 cm and <4 cm)
2. Histologically confirmed squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma
3. Planned for Type B or C radical hysterectomy
4. With adequate bone marrow, renal, and hepatic function

   * WBC >3.0 × 10⁹ cells/L
   * Platelets >100 × 10⁹ cells/L
   * Creatinine <180 μmol/L
   * Bilirubin <1.5 × normal range
   * AST, ALT < 3 × normal range
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
6. Previous history of other invasive malignancies with no evidence of recurrence for at least 5 years
7. Signed and approved consent form

II. Exclusion Criteria:

1. Histological types other than squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma
2. Tumor size less than 2 cm classified as 2018 FIGO stage IA1, IA2, or IB1 disease
3. The following are observed on preoperative CT or MRI

   * Tumor size ≥4 cm
   * Lymph node metastasis (short axis ≥15 mm)
   * Paracervical invasion
   * Bladder or rectal invasion
   * Distant metastasis
4. Prior pelvic or abdominal radiotherapy
5. Prior neoadjuvant chemotherapy before surgery
6. Unsuitable for surgery due to severe systemic disease at the investigator's discretion
7. Difficult to consider intraoperative lymphatic mapping due to

   * Allergy to triphenylmethane compounds
   * History of prior retroperitoneal surgery
   * History of prior pelvic radiotherapy
   * Cases where cold knife or loop electrosurgical excision procedure (LEEP) was performed within 4 weeks prior to study participation
   * Allergy to triphenylmethane compounds

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2034-12-31 (Estimated); Study Completion 2035-06-30 (Estimated)

PRIMARY OUTCOMES:
4.5-year progression-free survival rate | Up to 4.5 years after enrollment
  Proportion of patients alive without disease progression or death at 4.5 years after enrollment, as assessed by radiographic imaging and/or clinical criteria

SECONDARY OUTCOMES:
Intraoperative complcation rate | During surgery
  Proportion of patients experiencing intraoperative complications, including anesthesia-related adverse events, bleeding, organ injury, or other unexpected intraoperative events
Postoperative acute complication rate within 4 weeks | Within 4 weeks after surgery
  Proportion of patients experiencing acute postoperative complications within 4 weeks after surgery, including urinary tract infection, cardiopulmonary complications, thromboembolic events, bleeding or organ dysfunction
Postoperative complication rate after 4 weeks | Greater than 4 weeks up to 12 months post-surgery
  Proportion of patients experiencing acute postoperative complications after 4 weeks after surgery, including lymphedema, incisional hernia and dehiscence
Operation time | Peri-procedural
  The total duration of a surgical procedure, specifically measured from the initial surgical incision to the final closure of the wound
Estimated blood loss | Peri-procedural
  The approximated volume of blood a patient is believed to have lost during a surgical procedure or an injury.
Transfusion requirement | From the surgical incision to the end of surgery (skin closure)
  The need for administration of red blood cells to a patient to restore or maintain adequate oxygen-carrying capacity, hemostasis, and blood volume.
Length of hospitalization | From date of hospital admission to date of hospital discharge, assessed up to 30 days.
  The total duration (in days) between a patient's hospital admission and discharge.
Postoperative pain | Assessed at each visit from Visit 2 (2 weeks) and Visit 17 (54 months). The score can range from 0 to 10, with a higher score indicating more severe pain.
  Patient-reported pain intensity measured using a numeric rating scale (0-10)
Functional Assessment of Cancer Therapy-Cervix (FACT-Cx) | Assessed at Visit 1(within 4 weeks), Visit 3(2 weeks), Visit 4(6 weeks), Visit 5(3 months), Visit 6(6 months), Visit 10(18 months), Visit 13(30 months), Visit 17(54 months).
  Patient-reported quality of life evaluated using the FACT-Cx questionnaire, which includes physical, social/family, emotional, functional well-being, and cervix cancer-specific concerns. The FACT-Cx total score ranges from 0 to 168, with a higher score indicating better quality of life.
EQ-5D-5L | Assessed at Visit 1 (within 4 weeks), Visit 3 (2 weeks), Visit 4 (6 weeks), Visit 5 (3 months), Visit 6 (6 months). The score ranges from -0.594 to 1.000, showing that higher scores mean healthier.
  Patient-reported health-related quality of life assessed using the EQ-5D questionnaire, including five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Scores will be converted to index values based on country-specific value sets, and EQ visual analog scale (EQ-VAS) will also be recorded. Higher scores indicate better health status.
The 12-item Short Form Health Survey (SF-12) | Assessed at Visit 1 (within 4 weeks), Visit 3 (2 weeks), Visit 4 (6 weeks), Visit 5 (3 months), Visit 6 (6 months). The score can range from 0 to 100, with a higher score indicating less severe symptoms.
  Patient-reported health-related quality of life assessed using the SF-12 questionnaire, which yields Physical Component Summary (PCS) and Mental Component Summary (MCS) scores. Higher scores indicate better health status.
Pelvic Floor Distress Inventory (PFDI) | Assessed at Visit 1 (within 4 weeks), Visit 5 (3 months), Visit 6 (6 months), Visit 10 (18 months), Visit 13 (30 months), Visit 15 (42 months), Visit 17 (54 months). The score can range from 0 to 300, with a higher score indicating more severe symptoms.
  Patient-reported pelvic floor dysfunction symptoms assessed using the PFDI questionnaire, which includes subscales for urinary, colorectal-anal, and pelvic organ prolapse symptoms. Higher scores indicate greater symptom distress
4.5-year overall survival rate | Up to 4.5 years after surgery
  Overall survival defined as the time from date of surgery to death from any cause. The 4.5-year survival rate will be estimated using the Kaplan-Meier method. Patients alive at the end of follow-up will be censored at the last known contact.
Recurrence pattern at first recurrence | From date of surgery through 4.5 years postoperatively
  Distribution of first recurrence sites categorized as central, pelvic sidewall, and distant metastases. Recurrence must be radiologically or pathologically confirmed.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No